CLINICAL TRIAL: NCT02259946
Title: A Randomised, Double-blind, Placebo-controlled (Within Dose Groups) Study to Assess Safety, Tolerability and Pharmacokinetics of Single Rising Inhaled Doses (2.5 μg, 5 μg, 10 μg, 20 μg and 40 μg) of BI 1744 CL (Administered With the Respimat®) in Free Dose Combination With Tiotropium Bromide 5 μg ( for Doses up to and Including 20 μg BI 1744 CL), 10 μg (for Doses of 20 μg and 40 μg BI 1744 CL) (Administered With the Respimat®) in Healthy Male Volunteers
Brief Title: Study to Investigate Safety and Tolerability of BI 1744 CL in Free Dose Combination With Tiotropium Bromide Both Administered by Respimat® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.1
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — olodaterol; Tiotropium Bromide

ARMS (2):
- BI 1744 CL - single rising dose + Tiotropium (Experimental): Single rising dose of BI 1744 CL (conjointly with Tiotropium bromide)
  Interventions: Drug: BI 1744 CL; Drug: Tiotropium bromide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1744 CL
  Arms: BI 1744 CL - single rising dose + Tiotropium
Drug: Placebo
  Arms: Placebo
Drug: Tiotropium bromide
  Arms: BI 1744 CL - single rising dose + Tiotropium

SUMMARY:
Study to investigate safety and tolerability of single, inhaled doses (2.5 μg, 5 μg, 10 μg, 20 μg and 40 μg) of BI 1744 CL in free dose combination with tiotropium bromide 5 μg (for doses up to and including 20 μg BI 1744 CL) and 10 μg (for doses of 20 μg and 40 μg BI 1744 CL), both administered by Respimat® in healthy male volunteers. Also, to investigate the pharmacokinetics of BI 1744 BS and tiotropium bromide in such combinations, to explore their dose proportionality, and to explore the pharmacodynamic effects of the treatments on selected metabolic and respiratory parameters

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male based upon a complete medical history, including the physical examination, regarding vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead ECG measurement, and clinical laboratory tests. Absence of any clinically relevant abnormality. Absence of any clinically relevant concomitant disease
2. Age ≥21 and ≤50 years
3. BMI ≥18.5 and <30 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
2. Evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to randomization
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to enrolment in the study or during the study
10. Participation in another trial with an investigational drug within 2 months prior to randomization
11. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
12. Inability to refrain from smoking on trial days as judged by the investigator
13. Alcohol abuse (regularly more than 40 g alcohol per day for men)
14. Drug abuse
15. Blood donation (more than 100 mL blood within 4 weeks prior to randomisation or during the trial)
16. Excessive physical activities within 1 week prior to randomization or during the trial
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of the study centre

    Additionally, following exclusion criteria that are of particular relevance with regard to the known properties of BI 1744 CL as a ß-adrenoceptor agonist must be adhered to:
19. Asthma or history of pulmonary hyperreactivity
20. Hyperthyrosis
21. Allergic rhinitis in need of treatment
22. Clinically relevant cardiac arrhythmia
23. Paroxysmal tachycardia

    Furthermore, the following exclusion criteria that are of particular relevance with regard to the known properties of tiotropium as an antimuscarinic anticholinergic agent must be adhered to:
24. Hypersensitivity to tiotropium and/or related drugs of these classes
25. History of narrow-angle glaucoma
26. History of prostatic hyperplasia
27. History of bladder-neck obstruction

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-04; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal findings in physical examination | up to 12 days after drug administration
Number of participants with abnormal changes in laboratory parameters | up to 12 days after drug administration
Number of participants with clinically significant changes in vital signs | up to 12 days after drug administration
  blood pressure (BP), pulse rate (PR), respiratory rate (RR)
Number of participants with adverse events | up to 12 days after drug administration
Number of participants with clinically significant changes in 12-lead ECG | up to 12 days after drug administration
  cardiac axis, heart rate, PQ interval, QRS interval, uncorrected QT interval, HR-corrected QT-interval according to Bazett and Fridericia
Number of abnormal findings on oropharyngeal inspection | up to 24 hours after drug administration
Number of abnormal findings on pulmonary auscultation | up to 24 hours after drug administration
Assessment of tolerability by investigator on a 4-point scale | 12 days after drug administration
Change in Airway resistance (Raw) | up to 24 hours after drug administration
  measured by whole-body plethysmography
Change in specific conductance (sGaw) | up to 24 hours after drug administration
  measured by whole-body plethysmography
Change in Cyclic aminomonophosphate (cAMP) | up to 6 hours after drug administration
Change in potassium | up to 6 hours after drug administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of BI 1744 BS and tiotropium in plasma) | up to 96 hours after drug administration
tmax (time from dosing to maximum measured concentration) | up to 96 hours after drug administration
AUC0-∞ (area under the concentration-time curve of BI 1744 BS and tiotropium in plasma over the time interval from 0 extrapolated to infinity) | up to 96 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte salmeterol in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 96 hours after drug administration
%AUCtz-∞ (percentage of the extrapolated part of the total AUC0-∞) | up to 96 hours after drug administration
λz (terminal rate constant in plasma) | up to 96 hours after drug administration
t1/2 (terminal half-life of BI 1744 BS and tiotropium in plasma) | up to 96 hours after drug administration
MRTih (mean residence time of BI 1744 BS and tiotropium in the body after inhalation) | up to 96 hours after drug administration
CL/F (apparent clearance of BI 1744 BS and tiotropium in plasma after extravascular administration) | up to 96 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 96 hours after drug administration
Aet1-t2 (amount of BI 1744 BS and tiotropium eliminated in urine from the time point t1 to time point t2) | up to 96 hours after drug administration
fet1-t2 (fraction of BI 1744 BS and tiotropium eliminated in urine from time point t1 to time point t2) | up to 96 hours after drug administration
CLR,t1-t2 (renal clearance of BI 1744 BS and tiotropium from the time point t1 until the time point t2) | up to 96 hours after drug administration